CLINICAL TRIAL: NCT06013436
Title: Autologous Serum Tears Combined With 0.05% Cyclosporin Eye Drop Improve Corneal Nerve Density in Patients With Sjögren's Syndrome Dry Eye
Brief Title: AST Combined With 0.05% Cyclosporin Eye Drop Improve Corneal Nerve Density in Patients With SS Dry Eye
Acronym: AST/SS
Status: Completed | Type: Observational
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jiachun Hu, Resident physician, Chengdu University of Traditional Chinese Medicine
Other Study IDs: 22LLZX10
Record Dates: First submitted 2023-07-26; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Sjogren's Syndrome; Dry Eye; Ocular Surface Disease
Keywords: autologous serum tears; 0.05% cyclosporin eye drop; cornea nerves
MeSH Terms: conditions — Sjogren's Syndrome; Dry Eye Syndromes | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental group: Autologous serum tears, twelve times daily（per hour）, 12weeks. 0.05% cyclosporin eye drop, twice times daily, 12weeks.
  Interventions: Drug: Autologous serum tears combined with 0.05% cyclosporin eye drop

INTERVENTIONS:
Drug: Autologous serum tears combined with 0.05% cyclosporin eye drop — All patients administrated autologous serum tears twelve times daily（per hour） and 0.05% cyclosporin eye drop twice times daily in each eye for 12 weeks.
  Other Names: Ciclosporin Eye Drops(II)（Cyclone® ，SHENYANG XINGQI PHARMACEUTICAL Co., Ltd.）

SUMMARY:
The objective of the present study was to evaluate the efficacy of autologous serum tears combined with 0.05% cyclosporin eye drop in treating Sjögren's syndrome dry eye and their effect on corneal nerves. We assessed the impact of 12-week AST combined with 0.05% cyclosporin eye drop treatment on signs, symptoms, and sub-basal nerve density (SND) in patients with dry eyes related to Sjogren's syndrome.

DETAILED DESCRIPTION:
Objective: To describe the clinical efficacy and safety of the treatment of Sjögren's syndrome dry eye using autologous serum tears combined with 0.05% cyclosporin eye drop and to evaluate their effect on corneal nerves.

Design: Singal-center, prospective, observational study. Patients and methods: Thirty eyes of fifteen patients with dry eye related to Sjögren syndrome were enrolled in this study. Following a 4-week washout period, the treatment was inverted for each patient for the same duration and treatment. Ocular Surface Disease Index (OSDI), tear film, break-up time, corneal staining with the use of fluorescein, Schirmer's test and corneal confocal microscopy were investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients were diagnosed with SS according to the classification criteria defined by the American-European Consensus Group for the diagnosis of SS and also diagnosed with severe DED based on the consensus of Chinese dry eye experts.
* Age 18-65 years old.
* Controlled collagen disease by the same rheumatologists at least 3 months prior to the initiation of the trial.
* At least one eye that failed to respond to previous treatments including lartificial tears, topical ocular NSAIDs or corticosteroids.

Exclusion Criteria:

* Patients with DED related to meibomian gland dysfunction, blepharitis, abnormal blinking, conjunctival relaxation or any other diseases besides SS.
* Diagnosed with allergic conjunctivitis, uveitis, ocular hypertension, retinopathy and other eye diseases.
* Those who have a history of previous ocular oprations, eye injuries or contact lenses usage.
* Known hypersensitivity to experimental drugs or any of its ingredients.
* Necessity to modify the systemic treatment of previous diseases during the trial.
* Pregnancy or lactation.
* Severe systemic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From June 2022 to June 2023, moderate and severe dry eye patients with Sjogren's syndrome were treated in the Department of Ophthalmology and Rheumatology and Immunology of the Hospital of Chengdu University of Traditional Chinese Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
cornea nerves | 12 weeks
  cornea sub-basal nerve density
cornea staining score | 4 weeks
  to evaluate corneal epithelial repair（0= no staining; 1= less than 5 staining points; 2= more than 5 and less than 30 staining points within the range of two quadrants; and 3= staining exceeding two quadrants or staining points more than 30）

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | 4 weeks
  to assess the quality of life and clinical symptom；The survey generated a score ranging 0-100 (0 indicated absence of eye discomfort and 100 represented maximum eye discomfort)
Schirmer's test | 4 weeks
  to assess tear flow
tear film breakup time (TBUT) | 4 weeks
  to assess tear film stability

CONTACTS AND LOCATIONS:
Overall Officials: Jiachun Hu, Resident, Principal Investigator — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China